CLINICAL TRIAL: NCT00335725
Title: Multicentric Prospective, Randomised, Controlled Clinical Study on Clinical Efficacy and Tolerability of Urinary FSH (Fostimon® , IBSA) Versus r-FSH (Gonal-F®, Serono) in ICSI.
Brief Title: Efficacy and Tolerability of Human FSH Versus Recombinant FSH (Follitropin Alpha) in ICSI.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01GBF/FSH08
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Infertility
Keywords: Ovarian stimulation; Infertility; ICSI; FSH
MeSH Terms: conditions — Infertility | interventions — Follicle Stimulating Hormone; follitropin alfa

ARMS (2):
- Fostimon (Experimental): Fostimon is an highly purified FSH preparation.
  Interventions: Drug: Follicle Stimulating Hormone
- Gonal-F (Active Comparator): Gonal-F is a recombinant FSH preparation.
  Interventions: Drug: Follicle Stimulating Hormone

INTERVENTIONS:
Drug: Follicle Stimulating Hormone — subcutaneous injection of FSH. Starting dose: 225 IU.
  Other Names: highly purified human derived FSH; Fostimon
  Arms: Fostimon
Drug: Follicle Stimulating Hormone — subcutaneous injection of FSH. Starting dose: 225 IU.
  Other Names: rec FSH; Gonal F
  Arms: Gonal-F

SUMMARY:
Purpose of the study is the comparative evaluation of the clinical efficacy and of the general tolerability of two different subcutaneous FSH preparations (Fostimon® IBSA Vs Gonal-F® Serono) when administered in patients undergoing ICSI

DETAILED DESCRIPTION:
This is a multicentric, prospective, randomised, investigator blind, controlled clinical trial (phase III) of two parallel groups, one receiving the test drug FSH (Fostimon® , IBSA) and the other the reference drug FSH (Gonal-F®, Serono). The groups will be paired on the major prognostic criteria.

In effect, a double blind trial is not really feasible since the drugs presentations are very different. However, in IVF, drugs are usually dispensed and/or injected by a nurse and therefor the Investigator can be blind. Moreover, the used preparations will contain the same amount of gonadotrophin units (75 IU), will be repackaged in anonymous boxes and the following sentence will be written in the Patient Information Sheet: "You are required not to inform the Investigator about the product's name".

The randomisation is necessary to get groups as comparable as possible for all the other aspects. The multicentric design has the double interest of facilitating the patients' recruitment and of decreasing the biases related to attitudes in a specific centre.

ELIGIBILITY:
Inclusion Criteria:

Women undergoing ovarian stimulation for IntraCytoplasmic Sperm Injection (ICSI) with the following characteristics:

>/= 18 and < 40 years old BMI between 19 and 30 kg/m2 less than 3 previous completed cycles basal FSH level less than 10 IU/l within the 6 months prior to the study

Exclusion Criteria:

age < 18 and >/= 40 years primary ovarian failure or women known as poor responders, i.e. requiring more than 225 IU of FSH as starting dose in previous treatment cycles or having less than 3 oocytes retrieved or with an oestradiol serum concentration < 900 pmol/l (250 pg/ml) ovarian cysts > 20 mm oocyte donation thawed embryos replacement patients affected by pathologies associated with any contraindication of being pregnant ascertained or presumptive hypersensitivity to the active principle and/or their ingredients abnormal bleeding of undetermined origin uncontrolled thyroid or adrenal dysfunction neoplasias severe impairment of the renal and/or hepatic functions women deprived of their freedom by administrative or legal decision

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2003-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J G Grudzinskas, Prof, Principal Investigator — The Bridge Centre One St Thomas Street London Bridge London SE1 9RY, UK2.
Locations (7):
- France (6):
  - Private Consulting, Bron
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital Edouard Herriot, Lyon
  - Institut de Médecine de la Reproduction, Marseille
  - Hôpital Américain, Neuilly-sur-Seine
  - Hôpital Tenon, Paris
- Semmelweis Medical School, Budapest, Hungary

REFERENCES:
- [Background] GEMZELL CA, DICZFALUSY E, TILLINGER G. Clinical effect of human pituitary follicle-stimulating hormone (FSH). J Clin Endocrinol Metab. 1958 Dec;18(12):1333-48. doi: 10.1210/jcem-18-12-1333. No abstract available. PMID 13611018
- [Background] Thompson CR, Hansen LM. Pergonal (menotropins): a summary of clinical experience in the induction of ovulation and pregnancy. Fertil Steril. 1970 Dec;21(12):844-53. doi: 10.1016/s0015-0282(16)37925-0. No abstract available. PMID 5481991
- [Background] Oelsner G, Serr DM, Mashiach S, Blankstein J, Snyder M, Lunenfeld B. The study of induction of ovulation with menotropins: analysis of results of 1897 treatment cycles. Fertil Steril. 1978 Nov;30(5):538-44. doi: 10.1016/s0015-0282(16)43634-4. No abstract available. PMID 720642
- [Background] Schwartz M, Jewelewicz R, Dyrenfurth I, Tropper P, Vande Wiele RL. The use of human menopausal and chorionic gonadotropins for induction of ovulation. Sixteen years' experience at the Sloane Hospital for Women. Am J Obstet Gynecol. 1980 Dec 1;138(7 Pt 1):801-7. doi: 10.1016/s0002-9378(16)32740-5. PMID 6778212
- [Background] Notation AD, Tagatz GE, Steffes MW. Serum 17beta-estradiol. Index of follicular maturation during gonadotropin therapy. Obstet Gynecol. 1978 Feb;51(2):204-9. PMID 622235
- [Background] Dore PC, Rice C, Killick S. Human gonadotrophin preparations. May cause allergic reaction. BMJ. 1994 Jun 4;308(6942):1509. doi: 10.1136/bmj.308.6942.1509b. No abstract available. PMID 8019294
- [Background] Howles CM, Loumaye E, Giroud D, Luyet G. Multiple follicular development and ovarian steroidogenesis following subcutaneous administration of a highly purified urinary FSH preparation in pituitary desensitized women undergoing IVF: a multicentre European phase III study. Hum Reprod. 1994 Mar;9(3):424-30. doi: 10.1093/oxfordjournals.humrep.a138522. PMID 8006130
- [Background] Wikland M, Borg J, Hamberger L, Svalander P. Simplification of IVF: minimal monitoring and the use of subcutaneous highly purified FSH administration for ovulation induction. Hum Reprod. 1994 Aug;9(8):1430-6. doi: 10.1093/oxfordjournals.humrep.a138724. PMID 7989500
- [Background] Daya S, Gunby J. Recombinant versus urinary follicle stimulating hormone for ovarian stimulation in assisted reproduction. Hum Reprod. 1999 Sep;14(9):2207-15. doi: 10.1093/humrep/14.9.2207. PMID 10469682
- [Background] Remorgida V, Venturini PL, Anserini P, Lanera P, De Cecco L. Administration of pure follicle-stimulating hormone during gonadotropin-releasing hormone agonist therapy in patients with clomiphene-resistant polycystic ovarian disease: hormonal evaluations and clinical perspectives. Am J Obstet Gynecol. 1989 Jan;160(1):108-13. doi: 10.1016/0002-9378(89)90099-9. PMID 2492145
- [Background] Hackeloer BJ, Fleming R, Robinson HP, Adam AH, Coutts JR. Correlation of ultrasonic and endocrinologic assessment of human follicular development. Am J Obstet Gynecol. 1979 Sep 1;135(1):122-8. PMID 474642
- [Background] Venturoli S, Paradisi R, Fabbri R, Magrini O, Porcu E, Flamigni C. Comparison between human urinary follicle-stimulating hormone and human menopausal gonadotropin treatment in polycystic ovary. Obstet Gynecol. 1984 Jan;63(1):6-11. PMID 6419189
- [Background] Mendelson EB, Bohm-Velez M, Joseph N, Neiman HL. Gynecologic imaging: comparison of transabdominal and transvaginal sonography. Radiology. 1988 Feb;166(2):321-4. doi: 10.1148/radiology.166.2.3275976.
- [Background] Fleischer AC. Transabdominal and transvaginal sonography of ovarian masses. Clin Obstet Gynecol. 1991 Jun;34(2):433-42. doi: 10.1097/00003081-199106000-00027. PMID 1868645
- [Background] Wang CF, Gemzell C. The use of human gonadotropins for the induction of ovulation in women with polycystic ovarian disease. Fertil Steril. 1980 May;33(5):479-86. doi: 10.1016/s0015-0282(16)44711-4. PMID 6768596

RESULTS

PARTICIPANT FLOW:
Groups:
- Fostimon: Highly purified FSH
- Gonal-f: Recombinant FSH
Period: Overall Study
Arm/Group | Fostimon | Gonal-f
Started | 75 | 76
Completed | 71 | 71
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fostimon | Gonal-f | Total
Number analyzed (Participants) | 75 | 76 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (4.0) | 30.0 (3.6) | 30.0 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 76 | 151
  Male | 0 | 0 | 0
basal FSH [Mean (Standard Deviation); unit: IU/L] | 5.9 (2.5) | 6.0 (1.9) | 6.0 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Oocytes Retrieved
Description: Total number of oocytes retrieved
Time Frame: 10 days after stimulation start
Population: patients who started the stimulation with FSH
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Fostimon | Gonal-f
Number analyzed (Participants) | 73 | 72
oocytes | 10.9 (4.9) | 12.0 (5.6)

2. Secondary Outcome: Clinical Pregnancy Rate
Description: clinical pregnancy rate defined as the presence of gestation sac and heart beat.
Time Frame: 6 weeks after treatment start
Population: patients who started the FSH treatment
Measure: Number; unit: percentage of treated patients
Arm/Group | Fostimon | Gonal-F
Number analyzed (Participants) | 73 | 72
percentage of treated patients | 30.1 | 29.2

ADVERSE EVENTS:
Arm/Group | Fostimon | Gonal-F
Serious Adverse Events (participants affected / at risk) | 2/73 | 5/72
Other Adverse Events (participants affected / at risk) | 3/73 | 3/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fostimon (N=73) | Gonal-F (N=72)
OHSS (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (4)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fostimon (N=73) | Gonal-F (N=72)
spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Ovarian cyst (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
tiredness (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No